CLINICAL TRIAL: NCT02095626
Title: Pilot Study to Investigate the Clinical Effect of Orally Inhaled AP301 on Treatment of Primary Graft Dysfunction (PGD) in Mechanically Ventilated Patients After Primary Lung Transplantation
Brief Title: Study in Intensive Care Patients Regarding the Effect of Inhaled AP-301 After Primary Graft Dysfunction After Lung Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apeptico Forschung und Entwicklung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP-301-III-001; 2013-000716-21 (EudraCT Number)
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: PGD Primary Graft Dysfunction
Keywords: Peptide
MeSH Terms: interventions — AP301 peptide; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AP301 (Experimental): Treatment group
  Interventions: Drug: AP-301
- Saline solution (Placebo Comparator)
  Interventions: Drug: saline solution

INTERVENTIONS:
Drug: AP-301 — orally delivered doses of 87.6 mg AP301 (dose per subject, 5 ml nebulizer filling dose) are inhaled every 12 hours for a total of 7 days
  Arms: AP301
Drug: saline solution — placebo solution (0.9 % physiologic NaCl, 5 ml nebulizer filling dose) is inhaled every 12 hours for a total of 7 days
  Arms: Saline solution

SUMMARY:
The purpose of this study is to investigate the effect of orally inhaled AP-301 on primary graft dysfunction after lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Being a male or female recipient on the AKH's waiting list for primary single or double LuTX
* PGD score ≥ 1 within 72 hours after LuTX
* Informed consent is available

Exclusion Criteria:

* History of clinically relevant allergies or idiosyncrasies to AP301 or any other inactive ingredient(s) of the investigational product
* Postoperative ECMO support
* Paediatric /adolescent recipients (< 18 years)
* Lobar transplantation
* Retransplantation
* Combined solid organ transplants
* Participation in other drug trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
P/F ratio | 7 days
  The changes of the P/F ratio from T0 (time of PGD diagnosis) to day 7 of the treatment or to extubation of the patient

SECONDARY OUTCOMES:
EVLW | 7 days or until extubation
  Measurement of extravascular lung water

CONTACTS AND LOCATIONS:
Overall Officials: Walter Klepetko, Univ.Prof.Dr.med.univ., Principal Investigator — Medical University of Vienna
Locations (1):
- Division of Thoracic Surgery MedUni Vienna, Vienna, Austria